CLINICAL TRIAL: NCT01152216
Title: An Open-Label Extension of the CONCERT Protocol (DIM18) Evaluating Dimebon (Latrepirdine) in Patients With Alzheimer's Disease
Brief Title: An Extension of the CONCERT Protocol (DIM18)
Acronym: CONCERT PLUS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Medivation, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIM18EXT
Record Dates: First submitted 2010-06-25; First posted 2010-06-29 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — latrepirdine

ARMS (1):
- Dimebon (Experimental)
  Interventions: Drug: Dimebon

INTERVENTIONS:
Drug: Dimebon — 20 mg orally three times daily

SUMMARY:
An open-label extension study of the CONCERT (DIM18) protocol evaluating the safety of dimebon (latrepirdine) in subjects with With Mild-to-Moderate Alzheimer's Disease on Donepezil.

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of the 12 month DIM18 CONCERT study
* Mild-to-moderate Alzheimer's disease
* Probable AD, Diagnostic and Statistical Manual of Mental Disorders-IV-Text Revised (DSM-IV-TR)
* Mini-Mental State Exam (MMSE) score between 12 and 24, inclusive
* Stable on donepezil for at least 6 months

Exclusion Criteria:

* Other causes of dementia
* Major structural brain disease
* Unstable medical condition or significant hepatic or renal disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 672 (Actual)
Dates: Start 2010-04; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Safety | Through study discontinuation
  To evaluate the long-term safety and tolerability of dimebon (latrepirdine) in Alzheimer's disease (AD) patients who have completed 52 weeks of blinded treatment in the DIM18 (CONCERT) protocol.